CLINICAL TRIAL: NCT05644743
Title: Clinical Transformation of Organoid Model to Predict the Efficacy of GC in the Treatment of Intrahepatic Cholangiocarcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Chengjun Sui,MD (Other)
Responsible Party: Sponsor-Investigator, Chengjun Sui,MD, Deputy Director of the Special Needs Division, Eastern Hepatobiliary Surgery Hospital
Organization: Eastern Hepatobiliary Surgery Hospital (Other)
Other Study IDs: 202240313
Record Dates: First submitted 2022-11-30; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-11

CONDITIONS: Organoids; Intrahepatic Cholangiocarcinoma
Keywords: Organoid
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: gemcitabine + cisplatin — Gemcitabine intravenous drip, day 1, 8； Cisplatin intravenous drip, day 1； 3 weeks is a cycle, and 6 cycles are used continuously.

SUMMARY:
The clinical incidence of intrahepatic cholangiocarcinoma (ICC) is high and insidious, and the prognosis of advanced patients is poor. The clinical manifestations of traditional chemotherapy GC and emerging targeted therapy are different in most patients, and there is still no effective scheme to evaluate the differences in individual patient reactivity. Patient-derived tumor organoids (PDO) are 3D-cultured tissues based on tumor cell dryness that reproduce a variety of biological characteristics of parental tumors in vitro and have similar drug responsiveness to tumors in vivo. This project plans to use clinical cases and optimized organoid culture system to first construct relevant organoids from unresectable ICC patient puncture samples. Secondly, based on the organoid model of intrahepatic cholangiocarcinoma, the clinical efficacy of GC regimen was predicted, and in vitro and in vivo drug screening was conducted to explore the guidance of patient-derived tumor organoids for clinical treatment. Then, multi-omics data of organoids and in vitro and in vivo drug efficacy evaluation model were used to explore the drug resistance genes of intrahepatic cholangiocarcinoma, providing the basis for personalized drug screening and efficacy evaluation of intrahepatic cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

- Histologically confirmed intrahepatic cholangiocarcinoma They are between 18 and 80 years old Written informed and signed consent form Biopsy sample of the intrahepatic bile duct

Exclusion Criteria:

- Under 18, over 80 Informed consent cannot be given Biopsy samples were not available

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: All patients were histologically or cytologically diagnosed with locally advanced inoperable radical resectable or metastatic intrahepatic cholangiocarcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Consistency of organoids and clinical patient responses to drugs | 3 years
  A total of 20 unresectable ICC patients were selected and biopsies were performed before treatment to construct organoid models. All patients were treated with GC chemotherapy. Drug responses of organoids and clinical patients were compared to determine the feasibility of in vitro organoid culture as a drug screening platform. The samples of 3 patients who were sensitive to GC and 3 patients who were resistant to GC were sequenced to search for drug-resistant genes, and the differential drug-resistant genes were studied in vitro.
Construction of drug resistance prediction model | 3 years
  A total of 20 patients with advanced unresectable ICC were selected to verify whether they participated in drug resistance by combining 1-2 drug resistance genes previously screened and the currently recognized platinum-based drug resistance genes. The results were compared with those of organoid models to build an organoid-based drug resistance prediction model.

CONTACTS AND LOCATIONS:
Overall Officials: chengjun sui, dr., Principal Investigator — Deputy director

IPD SHARING:
Plan to Share IPD: Undecided
After the start of our research, we plan to share the data through the website to make more researchers know about our research.